CLINICAL TRIAL: NCT04000295
Title: AMELIE: A Phase 3 Randomized, Open-label, Multicenter Trial of Apatinib and Etoposide Capsule Versus Weekly Paclitaxel in Patients With Platinum Resistant or Refractory Ovarian Cancer
Brief Title: Apatinib and Etoposide Capsule Versus Weekly Paclitaxel in Patients With Platinum Resistant Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-OC-301
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — apatinib; Etoposide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib and Etoposide capsule (Experimental): Apatinib (375 mg qd, q3w) and Etoposide capsule(50 mg/d, d1-14, q3w) combination until disease progression or intolerable toxicity
  Interventions: Drug: Apatinib; Drug: Etoposide
- Weekly Paclitaxel (Active Comparator): Weekly Paclitaxel (80 mg/m2, d1, d8, d15, q3w) until disease progression or intolerable toxicity
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Apatinib — Subjects receive Apatinib orally, Dosage form: tablet, Strength: 375 mg/d
  Arms: Apatinib and Etoposide capsule
Drug: Etoposide — Subjects receive Etoposide capsule orally, d1-14, q3w, Dosage form: capsule, Strength: 50 mg/d
  Arms: Apatinib and Etoposide capsule
Drug: Paclitaxel — Subjects receive Weekly Paclitaxel, intravenously, d1, d8, d15, q3w, Dosage form: injectable, Strength: 80 mg/m2
  Arms: Weekly Paclitaxel

SUMMARY:
The study is conducted to evaluate the efficacy, safety and tolerability of apatinib (375 mg qd) and etoposide capsule (50 mg/d, d1-14, q3w) in subjects with platinum resistant or refractory ovarian cancer compared with weekly paclitaxel (80 mg/m2, d1, d8, d15, q3w).

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years and older
2. Epithelial ovarian, fallopian tube or primary peritoneal cancer
3. Platinum refractory and resistant disease (disease progression during platinum therapy or within 6 months of platinum therapy)
4. EOCG performance status of 0-1

Exclusion Criteria:

1. Uncontrolled hypertension ( systolic ≥140 mmHg or diastolic ≥90 mmHg despite antihypertensive therapy)
2. Known hypersensitivity to any of the study drugs or excipients.
3. Known hereditary or acquired bleeding and thrombotic tendencies (e.g. hemophiliacs, coagulation disorders, thrombocytopenia, etc.);
4. Congenital or acquired immune deficiency (e.g. HIV infected)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) by independent review committee(IRC) | up to approximately 2 years
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the IRC according to the RECIST criteria

SECONDARY OUTCOMES:
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | up to approximately 2 years
  Frequency and severity of Adverse Events or Serious Adverse Events as defined by CTCAE version 5.0
PFS by investigator | up to approximately 2 years
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigator according to the RECIST criteria
Objective Response Rate (ORR) | up to approximately 2 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed per RECIST 1.1 criteria as well as Gynecologic Cancer Intergroup (GCIG) cancer antigen (CA)-125 criteria.
Overall Survival (OS) | up to approximately 3 years
  OS is the time interval from the date of randomization to death from any cause.
EQ-5D-5L questionnaire | up to approximately 2 years
  EQ-5D-5L is a questionnaire that focus on issues specific to ovarian cancer.
FOSI-8 questionnaire | up to approximately 2 years
  FOSI-8 is a questionnaire that focus on issues specific to ovarian cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.